CLINICAL TRIAL: NCT02802254
Title: Increasing Risk Perception of Physical Activity Using Patient-targeted Feedback: Randomized Controlled Trial.
Brief Title: Increasing Risk Perception of Physical Activity Using Patient-targeted Feedback.
Acronym: RiskAct
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. Sebastian Kohlmann, Dr. rer. nat. Dipl. Psych., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1525/100
Record Dates: First submitted 2016-06-12; First posted 2016-06-16 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Hypertension; Coronary Disease; Cardiac Diseases
Keywords: physical activity; patient feedback; risk perception; pedometer
MeSH Terms: conditions — Hypertension; Coronary Disease; Heart Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pedometer+physical-activity-feedback (Experimental): At cardiac consultation patients receive a patient-targeted individual physical-activity-feedback.
  Interventions: Behavioral: Patient-targeted individual physical-activity-feedback; Device: Pedometer
- Pedometer-only (Active Comparator): Patients use a Pedometer in order to measure their daily step number
  Interventions: Device: Pedometer

INTERVENTIONS:
Behavioral: Patient-targeted individual physical-activity-feedback — At cardiac consultation receive an individual feedback on their personal physical activity level.
  Arms: Pedometer+physical-activity-feedback
Device: Pedometer — Patients receive a pedometer two weeks prior to cardiac consultation.

SUMMARY:
The aim of this study is to evaluate the efficiency of a minimal intervention on risk perception of physical inactivity in patients with known coronary heart disease (CHD) and patients at risk for CHD. Therefore half of the patients (intervention group) get a personal feedback on their individual level of physical activity measured by pedometers and self-report questionnaires plus information about the risk factor 'physical inactivity' for heart diseases. Following the hypotheses the feedback should increase the patients risk perception of physical inactivity and furthermore increase physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Known coronary heart disease or at least 2 risk factors for coronary heart disease
* Age: 18 years up to 75 years
* Sufficient language skills
* Access to a telephone
* Willingness to participate in telephone interviews
* "Informed consent"

Exclusion Criteria:

* Life threatening health status
* Severe somatic or/and psychological disorder that needs urgent treatment
* Hospital stay within the last 7 days
* Surgical intervention plus hospital stay for at least 3 days within the last 2 months
* Myocardial infarction within the last 3 month
* Musculoskeletal diseases, which have a strong influence on physical activity
* Severe cognitive or/and visual difficulties

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Risk perception of physical activity level | Outcome measure is assessed at one month follow-up
  time of measurement: one month after cardiac consultation

SECONDARY OUTCOMES:
Risk perception of physical activity level | Outcome measure is assessed at three months follow-up
  time of measurement: three months after cardiac consultation
Physical activity Level (Pedometer, time spent sitting, IPAQ) | Outcome measure is assessed at one month follow-up and three months follow-up
  time of measurement: one months and three months after cardiac consultation
Adherence to the pedometer | Outcome measure is assessed at one month follow-up and three months follow-up
  time of measurement: one months and three months after cardiac consultation
Satisfaction and acceptance of the feedback | Outcome measure is assessed at one month follow-up and three months follow-up
  time of measurement: one months and three months after cardiac consultation
Depression severity (PHQ-9) | Outcome measure is assessed at one month follow-up and three months follow-up
  time of measurement: one months and three months after cardiac consultation
Anxiety severity (GAD-7) | Outcome measure is assessed at one month follow-up and three months follow-up
  time of measurement: one months and three months after cardiac consultation
Somatic symptom severity (PHQ-15) | Outcome measure is assessed at one month follow-up and three months follow-up
  time of measurement: one months and three months after cardiac consultation
Quality of life (EQ-5D) | Outcome measure is assessed at one month follow-up and three months follow-up
  time of measurement: one months and three months after cardiac consultation
New York Heart Association Class | Outcome measure is assessed at one month follow-up and three months follow-up
  time of measurement: one months and three months after cardiac consultation
Canadian Cardiology Society Class | Outcome measure is assessed at one month follow-up and three months follow-up
  time of measurement: one months and three months after cardiac consultation

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Löwe, Prof. Dr., Study Director — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - University Heart Center, Medical Center Hamburg Eppendorf, Hamburg
  - Cardiologicum Hamburg, Hamburg

IPD SHARING:
Plan to Share IPD: No